CLINICAL TRIAL: NCT02331511
Title: Effect of Aspirin and Clopidogrel in Prevention of Venous Obstruction After Implantation of Cardiac Pacemaker and Defibrillator
Brief Title: Prevention of Venous Obstruction After Implantation of Cardiac Pacemaker and Defibrillator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Ali Akbarzadeh, Assistant proffesor of shahid beheshti university of medical sciences, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CVRC100
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Complication of Cardiac Defibrillator; Disorder of Cardiac Pacemaker System; Venous Occlusion
MeSH Terms: interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): No antiplatelet drug
  Interventions: Drug: placebo
- Aspirin (Active Comparator): Aspirin 80 mg daily
  Interventions: Drug: Aspirin 80 mg daily
- Clopidogrel (Active Comparator): Clopidogrel 75mg daily
  Interventions: Drug: Clopidogrel 75 mg daily

INTERVENTIONS:
Drug: placebo — placebo administration for 3 months after device(PPM,ICD,CRT) implantation
  Other Names: placebo 1 tablet daily
  Arms: placebo
Drug: Aspirin 80 mg daily — Aspirin 80 mg daily administration for 3 months after device(PPM,ICD,CRT) implantation
  Other Names: Aspirin
  Arms: Aspirin
Drug: Clopidogrel 75 mg daily — Clopidogrel administration for 3 months after device(PPM,ICD,CRT) implantation
  Other Names: Clopidogrel
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to determine whether Aspirin or Clopidogrel are effective in the prevention of venous obstruction after implantation of cardiac pacemaker or defibrillator.

DETAILED DESCRIPTION:
There are growing numbers of endocardial permanent pacemakers (PPM) and implantable cardioverter defibrillators (ICD) and cardiac resynchronization therapy (CRT) device. Asymptomatic obstruction of the access vein reported to have a high incidence (30-50%) in some studies. This complication can cause some difficulties in follow up procedures such as device upgrading. The purpose of this study is to determine whether Aspirin or Clopidogrel are effective in the prevention of venous obstruction after implantation of cardiac pacemaker or defibrillator.

ELIGIBILITY:
Inclusion Criteria:

* patients who referred for first implantation of pacemaker, implantable cardiac defibrillator, or cardiac re synchronization therapy device

Exclusion Criteria:

* history of malignancy
* history of coagulopathy or platelet disorder
* history of venous thromboembolism
* history of gastrointestinal hemorrhage or active gastroduodenal ulcer in past 6 months
* history of chronic kidney disorder or serum creatinine more than 1.5 mg/dl
* patients who are on anticoagulant or other antithrombotic drugs or who must be on dual antiplatelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Venus obstruction(axillary or subclavian vein) more than 50%(measure by venography) | 3 months

SECONDARY OUTCOMES:
major bleeding | 3 months
A composite of death of any cause, myocardial infarction, or cerebrovascular accident. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Saafi, M.D., Study Chair — Shahid Beheshti University of Medical Sciences; Mohammad Ali Akbarzadeh, M.D., Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid ModaressHospital, Tehran, Tehran Province, Iran